CLINICAL TRIAL: NCT03120923
Title: A Short Term Outcomes of Subacromial Injection of Combined Corticosteroid With Low Volume Compared to High Volume of Local Anesthetic for Rotator Cuff Impingement Syndrome: A Randomized Controlled Trials
Brief Title: Combined Corticosteroid With Low Volume Compared to High Volume in Impingement Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Jatupon Kongtharvonskul, Dr, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HE551338
Record Dates: First submitted 2017-04-16; First posted 2017-04-19 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Impingement Shoulder
Keywords: subacromial injection
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine 3 cc & Triamcinolone Acetonide (Experimental)
  Interventions: Drug: Lidocaine 3 cc; Drug: Triamcinolone Acetonide
- Lidocaine 9cc & Triamcinolone Acetonide (Active Comparator)
  Interventions: Drug: Lidocaine 9 cc; Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Lidocaine 3 cc
  Arms: Lidocaine 3 cc & Triamcinolone Acetonide
Drug: Lidocaine 9 cc — 9mL of 1% lidocaine plus 1mL of 40mg triamcinolone acetonide
  Arms: Lidocaine 9cc & Triamcinolone Acetonide
Drug: Triamcinolone Acetonide

SUMMARY:
This study aims to assess and compare the effectiveness of two different volumes of local anesthetic combined with 40mg of triamcinolone for subacromial injections in treating patients with rotator cuff impingement syndrome

DETAILED DESCRIPTION:
Patients with rotator cuff impingement syndrome were randomized to undergo subacromial injection with 10mL total volume of 1% lidocaine plus 40mg triamcinolone acetonide (n = 22), or a 4mL total volume of 1% lidocaine plus 40-mg triamcinolone acetonide (n = 23). Evaluations using a visual analog scale (VAS) for pain during motion, and the Western Ontario Rotator Cuff Index (WORC) were completed before treatment and 30 minutes, 2 weeks, and 8 weeks after injection.

ELIGIBILITY:
Inclusion Criteria:

1. participants with clinically diagnosed the rotator cuff impingement
2. participants aged 20 years and older
3. at least 1 month's duration
4. pain of moderate to severe intensity, defined as a score of 5 or more points on a 10-cm visual analog scale (VAS) rated from 0 (no pain) to 10 (worst imaginable pain)

Exclusion Criteria:

1. patients with adhesive capsulitis of the shoulder (normal radiograph of affected shoulder, and restriction of passive motion >30° in ≥2 planes of movement)
2. previous trauma history at currently affected shoulder
3. previous corticosteroid injection history at the affected shoulder
4. abnormal calcification and/or primary osteoarthritis of the shoulder joint on plain radiographs
5. use of medication such as antiplatelet agent or anticoagulation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
VAS | 8 weeks
  Visual analog score

SECONDARY OUTCOMES:
WORC | 8 weeks
  Western Ontario Rotator Cuff Index
Adverse reaction | 8 weeks

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boonard M, Sumanont S, Arirachakaran A, Apiwatanakul P, Boonrod A, Kanchanatawan W, Kongtharvonskul J. Short-term outcomes of subacromial injection of combined corticosteroid with low-volume compared to high-volume local anesthetic for rotator cuff impingement syndrome: a randomized controlled non-inferiority trial. Eur J Orthop Surg Traumatol. 2018 Aug;28(6):1079-1087. doi: 10.1007/s00590-018-2149-3. Epub 2018 Feb 8. PMID 29423865